CLINICAL TRIAL: NCT00902109
Title: Pilot Study to Compare the Humphrey Field Analyzer (HFA) 30-2 Swedish Interactive Threshold Algorithm (SITA) Standard Perimetry With the New Scotoma-Oriented Perimetry (SCOPE), Using a New Fast GATE (German Adaptive Threshold Estimation) in Glaucoma Patients Under Topic Therapy
Brief Title: Study to Compare Standard Perimetry With the New Scotoma-Oriented Perimetry (SCOPE) Using a New Fast German Adaptive Threshold Estimation (GATE) in Glaucoma Patients
Acronym: TRASCO
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital Tuebingen (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Principal Investigator, Ulrich Schiefer, Prof. Dr. med., University Hospital Tuebingen
Other Study IDs: SCOPE-G-BETA
Record Dates: First submitted 2009-05-12; First posted 2009-05-14 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2016-01

CONDITIONS: Primary Open Angle Glaucoma (POAG)
Keywords: visual field; perimetry; progression; POAG; glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle; Disease Progression; Glaucoma | interventions — Visual Field Tests; Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- perimetry, HRT, OCT: perimetry, HRT, OCT
  Interventions: Device: Perimetry; Device: Confocal Scanning Laser Tomography; Device: Optical Coherence Tomography (OCT)

INTERVENTIONS:
Device: Perimetry — different perimetric devices, different perimetric grids: Octopus: New Scotoma-Oriented Perimetry (SCOPE) Using a New Fast German Adaptive Threshold Estimation (GATE) HFA: 30-2, Sita (Swedish Interactive Thresholding Algorithm) full threshold
  Other Names: Humphrey Field Analyzer 745i (HFA), Interzeag Octopus 101
Device: Confocal Scanning Laser Tomography — HRT examinations for the clinical evaluation of the optic disc.
  Other Names: Heidelberg Retina Tomograph (HRT)
Device: Optical Coherence Tomography (OCT) — imaging of the retinal nerve fiber layer
  Other Names: Spectralis-OCT (Heidelberg Engineering, Heidelberg, Germany)

SUMMARY:
The purpose of this study is to compare the two psychophysical perimetric techniques regarding progression of the visual field.

ELIGIBILITY:
Inclusion Criteria:

* primary open angle glaucoma (POAG)
* spherical ametropia max. ± 8 dpt
* cylindrical ametropia max. ± 3 dpt
* distant visual acuity > 10/20
* pupil diameter > 3 mm

Exclusion Criteria:

* diabetic retinopathy
* asthma
* history of epilepsy or significant psychiatric disease
* medications known to effect visual field sensitivity
* infections (e.g., keratitis, conjunctivitis, uveitis)
* severe dry eyes
* miotic drug
* squint
* nystagmus
* albinism
* any ocular pathology, in either eye, that may interfere with the ability to obtain visual fields
* keratoconus
* intraocular surgery (except for uncomplicated cataract surgery) performed < 3 month prior to screening
* history or signs of any visual pathway affection other than glaucoma
* history or presence of macular disease and/or macular edema, ocular trauma, medications known to affect visual field sensitivity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: University Eye Hospital
Sampling Method: Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2010-04; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Comparison of rate of progression | 36 month
  Perimetric measures every 3 month over 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Schiefer, Prof. Dr. med., Principal Investigator — University Hospital Tuebingen
Locations (1):
- Institute for Ophthalmic Research, Tübingen, Germany

REFERENCES:
- [Background] Schiefer U, Pascual JP, Edmunds B, Feudner E, Hoffmann EM, Johnson CA, Lagreze WA, Pfeiffer N, Sample PA, Staubach F, Weleber RG, Vonthein R, Krapp E, Paetzold J. Comparison of the new perimetric GATE strategy with conventional full-threshold and SITA standard strategies. Invest Ophthalmol Vis Sci. 2009 Jan;50(1):488-94. doi: 10.1167/iovs.08-2229. Epub 2008 Dec 5. PMID 19060285